CLINICAL TRIAL: NCT06449612
Title: Telerehabilitation After a Stroke: Feasibility, Safety and Performance Evaluation of an Application Based Training Programme for Patients After a Stroke in the Subacute Phase
Brief Title: Feasibility, Safety and Performance Evaluation of an Application Based Training Programme for Patients After a Stroke
Acronym: TeleRehaStroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corina Schuster-Amft (Other)
Responsible Party: Sponsor-Investigator, Corina Schuster-Amft, Head of Research Department, Reha Rheinfelden
Organization: Reha Rheinfelden (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: TeleRehaStroke
Record Dates: First submitted 2024-05-27; First posted 2024-06-10 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Stroke
Keywords: Telerehabilitation; Stroke Rehabilitation; Exercise; Home-based Rehabilitation
MeSH Terms: conditions — Stroke; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 'TeleRehaStroke' Intervention Group (Experimental): The 'TeleRehaStroke' programme is an application-based training programme for patients after a stroke, comprising three main modules: (1) training, (2) coaching, and (3) monitoring:
  Training: Six-week training programmes have been created that focus on the lower extremity and balance. Via the application, patients are provided with a personalised training plan adapted to their individual impairments including exercise videos.
  Coaching: Participants will be accompanied by a coaching therapist via messenger, which is included in the application.
  Monitoring: Blood pressure measurements can be entered and saved in the application. Questionnaires can be sent to be filled in by the participants.
  Interventions: Device: TeleRehaStroke: Training programme using the 'Blended Clinic' mobile application

INTERVENTIONS:
Device: TeleRehaStroke: Training programme using the 'Blended Clinic' mobile application — Primary end users (patients after stroke) will be familiarised with the application and the 'TeleRehaStroke' programme in two to three sessions during their last two to three weeks prior to discharge from the inpatient rehabilitation centre. This includes performing daily exercises, wearing an activity tracker and measuring blood pressure daily. Following discharge from rehabilitation, they will continue to use the application for 12 weeks.
  Other Names: Blended Clinic, Blended Clinic AI, Nuremberg, Germany (https://blended.clinic/de/)

SUMMARY:
The goal of this investigation is to evaluate the feasibility, safety and performance of an application-based training programme in patients after a stroke in the subacute phase.

* Is the training programme 'TeleRehaStroke' using the mobile application 'Blended Clinic' for patients after a stroke feasible and usable?
* How is the user experience of the mobile application-based training programme?

Participants will:

* Get to know the programme and use the application 'Blended Clinic' during their last weeks before discharge from the inpatient rehabilitation.
* Be guided through inpatient setting, transition and outpatient setting and be accompanied by a coaching therapist via the application.
* Continue to use the application for 12 weeks after discharge from rehabilitation.

DETAILED DESCRIPTION:
It is challenging for patients after stroke to maintain motivation to continue and sustain training at home with the same intensity after an inpatient rehabilitation. An emerging approach is represented by digital applications that are easily and flexibly accessible from home. An existing virtual blended care environment 'Blended Clinic' (Blended Clinic AI GmbH) involves a mobile application that provides a training platform for patients after a stroke. The successor version 'TeleRehaStroke' builds on the previous version 'Strokecoach' that comprises three main modules: (1) training, (2) coaching, and (3) monitoring.

The aim of this evaluation is to assess feasibility, safety and performance of the 'TeleRehaStroke' programme for stroke patients in the transition phase from inpatient to outpatient rehabilitation.

Patients after a stroke will be recruited in the subacute phase. They will use the 'TeleRehaStroke' programme during their last weeks of their inpatient rehabilitation and for a further 12 weeks following their discharge to an outpatient setting. This includes daily exercises and blood pressure measurements. In addition, patients will receive coaching messages, educational content and questionnaires via the application. They will be accompanied by a coach via the app.

Feasibility outcomes, patient's descriptive, clinical- and performance-based parameters will be evaluated. Outcomes will be assessed at different time points.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Clinically confirmed stroke
* Modified Rankin Scale score 1-5
* Able, to read and understand German language
* Owns a smartphone or a tablet with stable internet connection and the operating system Android version 11 or iOS version 14 or higher

Exclusion Criteria:

* Severe Aphasia
* Clinically significant concomitant disease states: visual, neurological, cardiorespiratory, psychiatric, or orthopaedic limitations that prevent a participant from following the investigator's instructions or limit performance in an exercise programme
* Recent events such as surgery or other surgical procedures, fractures, which limit the performance in an exercise programme
* Known or suspected non-compliance, drug or alcohol abuse
* Participation in another investigation (with interventional therapy, investigational drug or another medical device) within the 30 days preceding and during the present investigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-07-26 (Actual); Primary Completion 2025-07-29 (Actual); Study Completion 2025-07-29 (Actual)

PRIMARY OUTCOMES:
Feasibility process-related parameters: Recruitment rate | through total study completion (up to 12 months)
  The number of screened patients versus included patients. It will be considered feasible if ≥40% of informed patients will be enrolled and ≥75% of targeted sample size will be reached.
Feasibility process-related parameters: Process evaluation | through total study completion (up to 12 months)
  The absolute duration of study-related duties of study personnel/coach in minutes during the inpatient and the outpatient period will be determined.
Feasibility of training-related parameters: (Serious) adverse events and device deficiencies | through study completion, up to 4 months
  Number of adverse events (i.e., deaths, serious and non-serious adverse events as well as device deficiencies) will be reported for each patient. The criterion for success is the incidence of an adverse event in <10% of participants.
Feasibility of training-related parameters: Acceptance | end of intervention, approx. after 4 months
  Patient satisfaction will be measured with the Net Promoter Score (NPS). It involves a single question ('How likely is it that you would recommend TeleRehaStroke to a friend or colleague?' with an 11-point rating scale. It will be considered as successful if the average satisfaction is ≥50%.
Feasibility of training-related parameters: Adherence to exercise and monitoring | through study completion, up to 4 months
  Exercise adherence will be measured as the ratio of completed versus planned trainings. Monitoring adherence will be measured as the ratio of completed versus planned blood pressure measurements and activity tracker wearing time. Adherence ≥70% will be considered as successful.
Feasibility of training-related parameters: Drop-out Rate | through total study completion (up to 12 months)
  It will be defined as successful if ≥80% of enrolled participants will complete the study.
Feasibility of mHealth-related parameters: Stability and maintenance | through total study completion (up to 12 months)
  The number and description of system errors will be determined and defined as acceptable if ≤3 system failures occur per week.
Feasibility of mHealth-related parameters: Usability measured with the System Usability Scale (SUS) | end of intervention, approx. after 4 months
  The SUS consists of 10 statements considering the system evaluated on a five-point rating scale from strongly agree to strongly disagree. Scores above 70 represent an acceptable usability, with scores smaller than 50 being judged as unacceptable.
Feasibility of mHealth-related parameters: Usability measured with the German version of mHealth App Usability Questionnaire (G-MAUQ) | end of intervention, approx. after 4 months
  The G-MAUQ consists of 18 items distributed across three dimensions: ease of use, interface and satisfaction and usefulness. Using a 7-point rating scale, from 1 (strongly agree) to 7 (strongly disagree), patients rate each item. An average scoring of ≥4 will count as successful.
Feasibility of mHealth-related parameters: Quality | end of intervention, approx. after 4 months
  The user version of the Quality Assessment of Health related Apps (AQUA) consists of 31 items and assesses seven basic dimension of app-quality. All items use a five-point rating scale from 5 (strongly agree) to 1 (strongly disagree). By calculating the mean score for each dimension, the quality of an app with regard to each of the dimensions can be determined and compared. By calculating the overall mean a total score can be determined. Success is defined if the average scoring in each dimension is ≥3.
Feasibility of mHealth-related parameters: Satisfaction | end of intervention, approx. after 4 months
  Patient's subjective satisfaction will be assessed using a visual analogue scale from not satisfied at all to extremely satisfied. ('How satisfied are you with the application?'). An average satisfaction of ≥50% is considered a success.
Feasibility of mHealth-related parameters: User- and training experience: | end of intervention, approx. after 4 months
  A self-designed feedback questionnaire with a five-point rating scale (1: extremely negative to 5: extremely positive) including specific questions related to user experience, interaction with the devices, and coaching experience will be used.
Feasibility of mHealth-related parameters: Perceived change | end of intervention, approx. after 4 months
  Patients' subjective global perceived change will be assessed using a visual analogue scale (VAS) from very much worse to very much improved ('How would you characterise the change?'). It will be considered as acceptable if the health status at least remains the same.

SECONDARY OUTCOMES:
Change in functional status as assessed by the Functional Independence Measure (FIM) | baseline, discharge (approx. 3 weeks), end of intervention (approx. 4 months)
  The FIM aims to evaluate the functional status of patients after a stroke throughout the rehabilitation process. It consists of 18 categories focusing on motor and cognitive function. Each category is rated on a 7-point rating scale (from 1: <25% independence to 7: 100% independence).
Change in ambulation as assessed by the Functional Ambulation Categories (FAC) | baseline, discharge (approx. 3 weeks), end of intervention (approx. 4 months)
  The FAC rates ambulation ability on a six-point rating scale from zero: unable to walk or assistance by walking through two or more assistants to 5: able to walk independently everywhere.
Cognition assessed by the Montreal Cognitive Assessment (MoCA) at baseline | baseline
  The MoCa consists of 30 items. The lowest possible score is zero, the highest is 30.
Level of impairment assessed by the National Institute of Health Stroke Scale (NIHSS) at baseline | baseline
  The NIHSS consists of 11 items, each item scored between zero and four, where zero indicates normal function of a specific ability, while a higher score indicates some level of impairment. The higher the total score, the severe the impairment caused by a stroke.
Change in disability level on the Modified Rankin Scale (mRS) | baseline, week 1, discharge (approx. week 3), week 10, end of intervention (approx. 4 months)
  The mRS measures the degree of disability or dependence in daily activities in patients after a stroke using a rating scale from zero (no symptoms at all) to six (dead). The mRS score will be evaluated by the study personnel or/and by the patients via the application.
Change in self-reported disability on the Stroke Impact Scale (SIS) | week 1, discharge (approx. week 3), week 10, end of intervention (approx. 4 months)
  The SIS is a self-report questionnaire that evaluates disability and health-related quality of life after stroke. The SIS consists of eight subscales (strength, hand function, mobility, activity of daily living, emotion, memory, communication and participation) comprising a total of 59 questions. Patients can rate each item in terms of difficulty on five-point rating scale (from 1: could not do at all to 5: not difficult at all). Final scores range from 0 to 100. The SIS includes an extra question on how much the patient feels that he/she has recovered from stroke that is rated on a scale from 0 to 100.
Change in health-related quality of life assessed by the 36-Item Short Form Healthy Survey (SF-36) | week 1, discharge (approx. week 3), week 10, end of intervention (approx. 4 months)
  The SF-36 consists of eight sections (physical functioning, role limitations due to physical problems, general health perceptions, vitality, social functioning, role limitation due to emotional problems, general mental health, and health transition) with eight scales scores, which are the weighted sums of the questions in their subscale (0 to 100). The lower the score the higher the impairment. Patients will fill out the questions via application.
Change in quality of life as assessed by the EuroQoL EQ-5D-3L | baseline, end of intervention (approx. 4 months)
  The EuroQoL consists of six questions about an individuals' quality of life in general, a visual analogue scale with a score from 0 to 100 and descriptive questions about five dimensions. Each dimension can be evaluated using a three-point rating scale (1: no problems, 2: some problems, 3: extreme problems). The descriptive system of the EQ-5D-3L produces a 5-digit health state profile, whereas the value sets are anchored on 11111 representing complete health.
Life-space mobility as assessed by the German Life-Space Assessment (LSA-G) | discharge (approx. week 3), week 10, end of intervention (approx. 4 months)
  The LSA-G consists of a questionnaire on five different life spaces: rooms besides the bedroom, area outside the house, neighbourhood, town or city lived in, outside of the town or city lived in. For each life space individuals are asked whether they visited these spaces and how often, whether they needed assistive devices or personal assistance. A life-space level can be determined as well as a composite score which ranges from 0 to 120 points (higher scores indicating better mobility).
Change in sitting balance as measured by the Trunk Impairment Scale (TIS) | baseline, end of intervention (approx. 4 months)
  The TIS assesses static (with three items) and dynamic (with four items, each repeated two or three times) sitting balance and trunk coordination (two items, each repeated twice) in sitting position in patients after a stroke . Score ranges from 0 to 23, where the higher score indicates better balance and coordination.
Change in mobility assessed by the Timed Up and Go (TUG) | baseline, end of intervention (approx. 4 months)
  The TUG is a clinical tool to assess mobility and the risk of falling. The time patients need to complete the task will be measured in seconds.
Blood pressure and heart rate | through study completion, up to 4 months
  Blood pressure and heart rate will be measured with a digital blood pressure measurement device (Medisana BU 510, medisana GmbH, Neuss, Germany).
Change in physical performance as assessed by the Short Physical Performance Battery (SPPB) | baseline, end of intervention (approx. 4 months)
  The SPPB is a group of measures that combines the results of gait speed, chair raise and balance tests. The scores range from 0 to 12 (0: worst performance; 12: best performance).
Physical activity - accelerometry | from start of the intervention to discharge (up to 3 weeks), and last 3 weeks before end of intervention (approx. after 3 months)
  Activity data will be assessed using the GENEActiv (Activinsights, Kimbolton, UK) activity tracker. Time (in min) spent in different activity levels and steps per day will be determined.

CONTACTS AND LOCATIONS:
Locations (1):
- Reha Rheinfelden, Rheinfelden, Canton of Aargau, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gaumann S, Ziller C, Paulissen N, Behrendt F, Suica Z, Cruts B, Gammerschlag L, Parmar K, Gerth HU, Bonati LH, Schuster-Amft C. START-the Swiss tele-assisted rehabilitation and training program to support transition from inpatient to outpatient care in the subacute phase after a stroke: feasibility, safety and performance evaluation. Front Digit Health. 2025 Jan 31;6:1496170. doi: 10.3389/fdgth.2024.1496170. eCollection 2024. PMID 39959919